CLINICAL TRIAL: NCT02141672
Title: A Randomized, Controlled Double-blind Study Comparing the Efficacy and Safety of Voclosporin (23.7 mg BID, or 39.5 mg BID) With Placebo in Achieving Remission in Patients With Active Lupus Nephritis
Brief Title: AURA-LV: Aurinia Urinary Protein Reduction Active - Lupus With Voclosporin (AURA-LV)
Acronym: AURA-LV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR-VCS-2012-01
Record Dates: First submitted 2014-05-14; First posted 2014-05-19 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; calcineurin inhibitors; voclosporin
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Voclosporin Low Dose (Experimental): Voclosporin, oral, 23.7 mg BID
  Interventions: Drug: Voclosporin Low Dose
- Voclosporin High Dose (Experimental): Voclosporin, oral 23.7 mg BID until Week 2, then voclosporin, oral, 39.5 mg BID
  Interventions: Drug: Voclosporin High Dose
- Placebo (Placebo Comparator): Low dose: Voclosporin placebo, oral, 3 capsules BID
  High dose: Voclosporin placebo, oral, 3 capsules BID until Week 2 then voclosporin placebo, oral, 5 capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voclosporin High Dose
  Other Names: ISA247
  Arms: Voclosporin High Dose
Drug: Voclosporin Low Dose
  Other Names: ISA247
  Arms: Voclosporin Low Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy of 2 doses of voclosporin compared to placebo in achieving complete remission after 24 weeks of therapy in subjects with active lupus nephritis.

DETAILED DESCRIPTION:
Voclosporin is a next generation CNI intended for use in the prevention of organ graft rejection and for the treatment of autoimmune diseases. The aim of the current study is to investigate whether voclosporin added to the standard of care treatment in active LN is able to reduce disease activity, as measured by a reduction in proteinuria. Two doses of voclosporin will be studied and compared in a placebo controlled trial on a background of MMF and corticosteroids. Patients with active, flaring LN will be eligible to enter the study. They are required to have a diagnosis of LN according to established diagnostic criteria (American College of Rheumatology) and clinical and biopsy features suggestive of active nephritis. Efficacy will be assessed by the ability of the drug combination to reduce the level of proteinuria while demonstrating an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects aged 18 to 75 years.

Diagnosis of systemic lupus erythematosus (SLE) according to the American College of Rheumatology criteria.

Kidney biopsy within 6 months prior to Screening (Visit 1) with a histologic diagnosis of lupus nephritis (International Society of Nephrology/Renal Pathology Society 2003 classification of lupus nephritis) Classes III, IV-S or IV-G, (A) or (A/C); or Class V, alone or in combination with Class III or IV.

Laboratory evidence of active nephritis at screening, defined as:

* Class III, IV-S or IV-G: Confirmed proteinuria ≥1,500 mg/24 hours when assessed by 24 hour urine collection, defined by a UPCR of ≥1.5 mg/mg assessed in a first morning void urine specimen (2 samples).
* Class V (alone or in combination with Class III or IV): Confirmed proteinuria ≥2,000 mg/24 hours when assessed by 24 hour urine collection, defined by a UPCR of ≥2 mg/mg assessed in a first morning void urine specimen (2 samples).

Exclusion Criteria:

Estimated glomerular filtration rate (eGFR) as calculated by the Chronic Kidney Disease Epidemiology Collaboration equation of ≤45 mL/min/1.73 m2.

Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.

A previous kidney transplant or planned transplant within study treatment period.

In the opinion of the Investigator, subject does not require long-term immunosuppressive treatment (in addition to corticosteroids).

Current or medical history of:

* Pancreatitis or gastrointestinal hemorrhage within 6 months prior to screening.
* Active unhealed peptic ulcer within 3 months prior to screening. If an ulcer has healed and the subject is on adequate therapy, the subject may be randomized.
* Congenital or acquired immunodeficiency.
* Clinically significant drug or alcohol abuse 2 years prior to screening.
* Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision. Subjects with cervical dysplasia that is cervical intraepithelial neoplasia 1, but have been treated with conization or loop electrosurgical excision procedure, and have had a normal repeat PAP are allowed.
* Lymphoproliferative disease or previous total lymphoid irradiation.
* Severe viral infection (such as CMV, HBV, HCV) within 3 months of screening; or known human immunodeficiency virus infection.
* Active tuberculosis (TB), or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid.

Other known clinically significant active medical conditions, such as:

* Severe cardiovascular disease including congestive heart failure, history of cardiac dysrhythmia or congenital long QT syndrome.
* Liver dysfunction (aspartate aminotransferase, alanine aminotransferase, or bilirubin greater than 2.5 times the upper limit of normal) at screening and confirmed before randomization.
* Chronic obstructive pulmonary disease or asthma requiring oral steroids.
* Bone marrow insufficiency unrelated to active SLE (according to Investigator judgment) with white blood cell count <2,500/mm3; absolute neutrophil count <1.3 x 103/μL; thrombocytopenia (platelet count <50,000/mm3).
* Active bleeding disorders.
* Current infection requiring IV antibiotics.

Any overlapping autoimmune condition for which the condition or the treatment of the condition may affect the study assessments or outcomes. Overlapping conditions for which the condition or treatment is not expected to affect assessments or outcomes are not excluded.

Subjects who are pregnant, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Anne Dooley, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (71):
- United States (14):
  - AURA-LV Site, Los Angeles, California
  - AURA-LV Site, Palo Alto, California
  - AURA-LV Site, Gainesville, Florida
  - AURA-LV Site, Miami, Florida
  - AURA-LV Site, Farmington Hills, Michigan
  - AURA-LV Site, Brooklyn, New York
  - AURA-LV Site, New York, New York
  - AURA-LV Site, Chapel Hill, North Carolina
  - AURA-LV Site, Charlotte, North Carolina
  - AURA-LV Site, Columbus, Ohio
  - AURA-LV Site, Hershey, Pennsylvania
  - AURA-LV Site, Chattanooga, Tennessee
  - AURA-LV Site, Dallas, Texas
  - AURA-LV Site, Houston, Texas
- AURA-LV Site, Dhaka, Bangladesh
- Belarus (2):
  - AURA-LV Site, Minsk
  - AURA-LV Site, Vitebsk
- Bulgaria (3):
  - AURA-L Site, Plovdiv
  - AURA-LV Site, Sofia
  - AURA-LV Site, Varna
- AURA-LV Site, Hong Kong, China
- Ecuador (2):
  - AURA-LV Site, Guayaquil
  - AURA-LV Site, Quito
- AURA-LV Site, Tbilisi, Georgia
- AURA-LV Site, Guatemala City, Guatemala
- Mexico (4):
  - AURA-LV Site, Guadalajara
  - AURA-LV Site, Mexicali
  - AURA-LV Site, Oaxaca City
  - AURA-LV Site, Tlalpan
- Philippines (6):
  - AURA-LV Site, Angeles City
  - AURA-LV Site, Batangas
  - AURA-LV Site, Cebu City
  - AURA-LV Site, Davao City
  - AURA-LV Site, Manila
  - AURA-LV Site, Quezon City
- Poland (4):
  - AURA-LV Site, Katowice
  - AURA-LV Site, Radom
  - AURA-LV Site, Warsaw
  - AURA-LV Site, Wroclaw
- Russia (11):
  - AURA-LV Site, Kazan'
  - AURA-LV Site, Kemerovo
  - AURA-LV Site, Moscow
  - AURA-LV Site, Omsk
  - AURA-LV Site, Orenburg
  - AURA-LV Site, Petrozavodsk
  - AURA-LV Site, Rostov-on-Don
  - AURA-LV Site, Saint Petersburg
  - AURA-LV Site, Saratov
  - AURA-LV Site, Tolyatti
  - AURA-LV Site, Yaroslavl
- Serbia (2):
  - AURA-LV Site, Belgrade
  - AURA-LV Site, Niš
- AURA-LV Site, Singapore, Singapore
- South Korea (4):
  - AURA-LV Site, Busan
  - AURA -LV Site, Daegu
  - AURA-LV Site, Seoul
  - AURA-LV Site, Wŏnju
- Spain (2):
  - AURA-LV Site, Barcelona
  - AURA-LV, Madrid
- Sri Lanka (4):
  - AURA-LV Site, Colombo
  - AUR-LV Site, Kandy
  - AURA-LV Site, Nugegoda
  - AURA-LV Site, Ragama
- Taiwan (2):
  - AURA-LV Site, Kaohsiung City
  - AURA-LV Site, Taoyuan
- Thailand (2):
  - AURA-LV Site, Bangkok
  - AURA-LV Site, Chiang Mai
- Ukraine (4):
  - AURA-LV Site, Kharkiv
  - AURA-LV Site, Kyiv
  - AURA-LV Site, Lutsk
  - AURA-LV Site, Zaporizhzhya

REFERENCES:
- [Background] Dooley MA, Jayne D, Ginzler EM, Isenberg D, Olsen NJ, Wofsy D, Eitner F, Appel GB, Contreras G, Lisk L, Solomons N; ALMS Group. Mycophenolate versus azathioprine as maintenance therapy for lupus nephritis. N Engl J Med. 2011 Nov 17;365(20):1886-95. doi: 10.1056/NEJMoa1014460. PMID 22087680
- [Background] Appel GB, Contreras G, Dooley MA, Ginzler EM, Isenberg D, Jayne D, Li LS, Mysler E, Sanchez-Guerrero J, Solomons N, Wofsy D; Aspreva Lupus Management Study Group. Mycophenolate mofetil versus cyclophosphamide for induction treatment of lupus nephritis. J Am Soc Nephrol. 2009 May;20(5):1103-12. doi: 10.1681/ASN.2008101028. Epub 2009 Apr 15. PMID 19369404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects were randomized in a ratio of 1:1:1 to receive either voclosporin 23.7 mg BID or 39.5 mg BID, or matching placebo for 48 weeks. All subjects were also to receive 2 g/day MMF. In addition, all subjects were to receive 0.5 g/day IV methylprednisolone on Days 1 and 2 before changing to a reducing course of oral corticosteroid therapy on Day 3.
Groups:
- Voclosporin Low Dose: Voclosporin oral 23.7 mg (3 capsules) BID
- Voclosporin High Dose: Voclosporin oral 23.7 mg BID until week 2 followed by 39.5 mg (5 capsules) BID
- Placebo: Placebo capsules matched to high dose or low dose voclosporin regimen.
Period: Overall Study
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Started | 89 | 88 | 88
Completed | 73 | 80 | 70
Not Completed | 16 | 8 | 18
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 10 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Physician Decision | 1 | 2 | 5
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 5
Not completed — refused to follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo | Total
Number analyzed (Participants) | 89 | 88 | 88 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (11.78) | 30.6 (9.59) | 33.1 (10.03) | 31.7 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 81 | 73 | 230
  Male | 13 | 7 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 13 | 35
  Not Hispanic or Latino | 80 | 75 | 75 | 230
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 3 | 9
  Asian | 52 | 44 | 36 | 132
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 6 | 5 | 14
  White | 30 | 36 | 42 | 108
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 6 | 21
  Bangladesh | 17 | 16 | 13 | 46
  Belarus | 1 | 8 | 4 | 13
  Bulgaria | 2 | 1 | 2 | 5
  Ecuador | 2 | 1 | 2 | 5
  Georgia | 1 | 1 | 3 | 5
  Guatemala | 2 | 6 | 3 | 11
  Hong Kong | 0 | 0 | 1 | 1
  South Korea | 3 | 2 | 2 | 7
  Mexico | 3 | 3 | 8 | 14
  Philippines | 20 | 13 | 10 | 43
  Poland | 2 | 0 | 2 | 4
  Russia | 10 | 9 | 13 | 32
  Serbia | 4 | 1 | 7 | 12
  Singapore | 0 | 1 | 0 | 1
  Spain | 1 | 0 | 0 | 1
  Sri Lanka | 5 | 4 | 5 | 14
  Taiwan | 2 | 1 | 2 | 5
  Thailand | 5 | 6 | 2 | 13
  Ukraine | 4 | 5 | 3 | 12
Lupus Nephritis history [Mean (Standard Deviation); unit: years]
  Years since diagnosis of LN (years) | 4.2 (5.14) | 3.2 (4.36) | 3.5 (4.03) | 3.7 (4.54)
  Years since first significant proteinuria (years) | 4.5 (5.53) | 3.3 (4.22) | 3.6 (4.06) | 3.8 (4.66)
Lupus Nephritis history - Baseline UPCR [Median (Standard Deviation); unit: mg/mg] | 5.16 (4.15) | 4.48 (3.03) | 4.43 (3.58) | 4.69 (3.6)
Lupus Nephritis history - Baseline eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m2] | 95.3 (28.4) | 104 (27.3) | 100.2 (27.05) | 99.8 (27.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Complete Renal Remission at 24 Weeks
Description: Complete remission is defined as:
  * Confirmed protein/creatinine ratio of ≤0.5 mg/mg and
  * eGFR ≥60 mL/min/1.73m2 or no confirmed decrease from baseline in eGFR of ≥20%. Subjects who received rescue medication for lupus nephritis or >10 mg prednisone for >3 consecutive days or >7 days total from 56 days prior to remission assessment until the time of the remission assessment were considered not achieving complete remission.
Time Frame: week 24
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants
  Achieved response | 29 | 24 | 17
  Did not achieve response | 60 | 64 | 71
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Voclosporin low dose vs. placebo; Test type: Superiority; p = 0.045, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.01 to 4.05]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p = 0.204, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.78 to 3.27]

2. Secondary Outcome: Number of Subjects Achieving Complete Renal Remission at 48 Weeks
Description: as for outcome 1
Time Frame: Week 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants
  Achieved response | 44 | 35 | 21
  Did not achieve response | 45 | 53 | 67
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Voclosporin low dose vs. placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.21, 95% CI 2-sided [1.68 to 6.13]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p = 0.026, Regression, Logistic; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.09 to 4.02]

3. Secondary Outcome: Number of Subjects Achieving Complete Renal Remission at 24 and 48 Weeks in the Presence of Low Dose Steroids
Description: Complete remission is defined as:
  * Confirmed protein/creatinine ratio of ≤0.5 mg/mg and
  * eGFR ≥60 mL/min/1.73m2 or no confirmed decrease from baseline in eGFR of ≥20%. Subjects who received rescue medication for lupus nephritis or >10 mg prednisone for >3 consecutive days or >7 days total from 56 days prior to remission assessment until the time of the remission assessment were considered not achieving complete remission.
  Low-dose steroids is defined as use of ≤5 mg prednisone for 8 weeks leading up to the Week 24 visit date or for 12 weeks leading up to the Week 48 visit date.
Time Frame: Weeks 24 and 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants
  Achieved response at week 24 | 26 | 23 | 17
  Achieved response at week 48 | 29 | 26 | 18
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Test type: Superiority; p = 0.066, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI 2-sided [0.96 to 3.78]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Test type: Superiority; p = 0.162, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.82 to 3.28]

4. Secondary Outcome: Time to Complete Remission (Number of Weeks)
Description: Time to Complete Remission is defined as time from first dose of voclosporin/placebo to UPCR ≤ 0.5mg in the absence of rescue medication.
Time Frame: week 48
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
weeks | 19.7 [16.1 to 36.1] | 23.4 [13.7 to 33.4] | NA [48.1 to NA] — NA = insufficient number of participants with events
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Voclosporin low dose vs. placebo; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.26, 95% CI 2-sided [1.45 to 3.51]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.25, 95% CI 2-sided [1.46 to 3.47]

5. Secondary Outcome: Time to Sustained Early Complete Remission (Number of Weeks)
Description: Time to Sustained Complete Remission is defined as time from first dose of voclosporin/placebo to UPCR ≤ 0.5mg occurring at week 24 or earlier and sustained until week 48 in the absence of rescue medication.
Time Frame: week 48
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
weeks | NA [20.0 to NA] — NA = insufficient number of participants with events | NA [NA to NA] — NA = insufficient number of participants with events | NA [NA to NA] — NA = insufficient number of participants with events
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.89, 95% CI 2-sided [1.58 to 5.29]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p < 0.248, Regression, Cox; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [0.77 to 2.86]

6. Secondary Outcome: Number of Subjects Achieving Sustained Early Complete Remission
Description: Sustained early complete remission defined as complete remission that occurred on or before Week 24 and was sustained through Week 48
Time Frame: week 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants | 36 | 22 | 15

7. Secondary Outcome: Time to Partial Remission (Number of Weeks)
Description: Time to partial Remission is defined as time from first dose of voclosporin/placebo to 50% UPCR reduction sustained until week 48 in the absence of rescue medication.
Time Frame: week 48
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
weeks | 4.3 [2.6 to 5.9] | 4.4 [4.1 to 6.1] | 6.6 [4.6 to 8.6]
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Test type: Superiority; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 1.63, 95% CI 2-sided [1.16 to 2.27]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [1.25 to 2.43]

8. Secondary Outcome: Number of Subjects Achieving Partial Remission
Description: Partial remission is defined as a 50% reduction in UPCR from baseline at Week 24 and Week 48.
Time Frame: week 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants | 76 | 82 | 67

9. Secondary Outcome: Number of Subjects Achieving, and Remaining in, Complete Remission
Description: Sustained complete remission defined as the first occurrence of complete remission that was sustained through Week 48
Time Frame: week 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants
  Number of Participants Achieving Complete Remission | 57 | 61 | 32
  Number of Participants Remaining in Complete Remission | 19 | 28 | 10
  Number of Participants with Second Increase of UPCR >0.5 mg/mg | 38 | 33 | 22
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Voclosporin low dose vs. placebo; Test type: Superiority; p = 0.980, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.45 to 2.15]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p = 0.118, Regression, Cox; Hazard Ratio (HR) = 1.98, 95% CI 2-sided [0.95 to 4.16]

10. Secondary Outcome: Duration of Complete Remission (Number of Weeks)
Description: Duration of Complete Remission is defined as time of first occurrence of UPCR ≤ 0.5 mg/mg until the second increase above 0.5 mg/mg (i.e. a single occurrence above 0.5 is permitted) or use of rescue medication.
Time Frame: week 48
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
weeks | 49 [42.1 to 49.0] | 25 [23.3 to NA] — NA = insufficient number of participants with events | NA [26.3 to NA] — NA = insufficient number of participants with events

11. Secondary Outcome: Number of Subjects Achieving Partial Renal Remission at 24 and 48 Weeks
Description: Number of patients with partial Remission is defined as time from first dose of voclosporin/placebo to 50% UPCR reduction at week 24 or week 48 in the absence of rescue medication.
Time Frame: week 24 and 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants
  Achieved partial remission at week 24 | 62 | 58 | 43
  Achieved partial remission at week 48 | 61 | 63 | 42
Statistical Analysis 1: Comparison: Voclosporin Low Dose; week 24; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.26 to 4.33]
Statistical Analysis 2: Comparison: Voclosporin High Dose; week 24; Test type: Superiority; p = 0.024, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.1 to 3.76]
Statistical Analysis 3: Comparison: Voclosporin Low Dose; week 48; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.27 to 4.33]
Statistical Analysis 4: Comparison: Voclosporin High Dose; week 48; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.43 to 5.02]

12. Secondary Outcome: Time to Sustained Partial Remission (Number of Weeks)
Description: Time to sustained partial Remission is defined as time from first dose of voclosporin/placebo to 50% UPCR reduction sustained until week 48 in the absence of rescue medication.
Time Frame: week 48
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
weeks | 6.3 [4.0 to 11.9] | 8.1 [6.1 to 16.6] | 26.9 [16.1 to NA] — NA = insufficient number of participants with events
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Voclosporin low dose vs. placebo; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.03, 95% CI 2-sided [1.36 to 3.03]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 1.81, 95% CI 2-sided [1.22 to 2.69]

13. Secondary Outcome: Number of Subjects Achieving Sustained Partial Remission
Description: Sustained partial remission defined as the first occurrence of partial remission that was sustained through Week 48
Time Frame: week 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants | 61 | 63 | 42

14. Secondary Outcome: Time to Sustained Early Partial Remission (Number of Weeks)
Description: Time to sustained early partial Remission is defined as time from first dose of voclosporin/placebo to 50% UPCR reduction occurring at week 24 or earlier and sustained until week 48 in the absence of rescue medication.
Time Frame: week 48
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
weeks | 6.3 [4.0 to 11.9] | 8.1 [6.1 to 16.6] | NA [16.1 to NA] — NA = insufficient number of participants with events
Statistical Analysis 1: Comparison: Voclosporin Low Dose; Voclosporin low dose vs. placebo; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 2.21, 95% CI 2-sided [1.45 to 3.36]
Statistical Analysis 2: Comparison: Voclosporin High Dose; Voclosporin high dose vs. placebo; Test type: Superiority; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 1.87, 95% CI 2-sided [1.23 to 2.84]

15. Secondary Outcome: Number of Subjects Achieving Sustained Early Partial Remission
Description: Early partial remission defined as partial remission that occurred on or before Week 24 and was sustained through Week 48
Time Frame: week 48
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
Participants | 60 | 58 | 36

16. Secondary Outcome: Change From Baseline in UPCR at Weeks 24 and 48
Description: Change from baseline in urine protein creatinine ratio at weeks 24 and 48
Time Frame: Baseline, Week 24 and Week 48
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
mg/mg
  Baseline UPCR | 5.161 (4.151) | 4.476 (3.029) | 4.433 (3.58)
  week 24 UPCR | 1.021 (1.2369) | 1.356 (1.5204) | 2.266 (2.8534)
  CFB at week 24 | -3.769 (3.351) | -2.792 (2.6207) | -2.216 (3.9284)
  week 48 UPCR | 0.689 (0.9172) | 1.101 (1.3835) | 1.763 (1.9927)
  CFB at week 48 | -3.998 (3.4208) | -2.993 (2.6608) | -2.384 (3.454)

17. Secondary Outcome: Change From Baseline in Safety of Estrogens in Systemic Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) Score
Description: The SELENA-SLEDAI assesses disease activity within the last 10 days. Twenty-four items are scored for nine organ systems, and summed to a maximum of 105 points. A score of 6 is considered clinically significant and indicates active disease. For analysis purposes, a score ≥6 was categorized as "high". The 24 items are as follows: seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, hematuria, proteinuria, pyuria, new rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, increased DNA binding, fever, thrombocytopenia, and leukopenia.
Time Frame: Baseline, Week 24 and Week 48
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
Number analyzed (Participants) | 89 | 88 | 88
score on a scale
  SELENA-SLEDAI Score at baseline | 12.7 (6.37) | 13.9 (6.51) | 12.9 (6.57)
  SELENA-SLEDAI Score at week 24 | 6.2 (4.53) | 6.5 (5.42) | 8.8 (5.43)
  SELENA-SLEDAI Score change from baseline at week 24 | -6.3 (5.86) | -7.1 (7.41) | -4.5 (7.09)
  SELENA-SLEDAI Score at week 48 | 4.7 (5.06) | 5.3 (3.97) | 7.8 (5.93)
  SELENA-SLEDAI Score Change from baseline at week 48 | -7.9 (6.39) | -8.3 (6.93) | -5.3 (6.85)

ADVERSE EVENTS:
Time Frame: Week 52
Description: Treatment emergent AEs. Reporting period is from first dose up to 30 days after study completion or withdrawal
Arm/Group | Voclosporin Low Dose | Voclosporin High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 10/89 | 2/88 | 1/88
Serious Adverse Events (participants affected / at risk) | 25/89 | 22/88 | 14/88
Other Adverse Events (participants affected / at risk) | 82/89 | 85/88 | 75/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voclosporin Low Dose (N=89) | Voclosporin High Dose (N=88) | Placebo (N=88)
Pneumonia (Infections and infestations) | 5 | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 2 | 1
Sepsis (Infections and infestations) | 1 | 2 | 0
Body Tinea (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Herpes Zoster (Infections and infestations) | 0 | 1 | 1
Bacterial Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous Abcess (Infections and infestations) | 0 | 1 | 0
Tuberculosis of Genitourinary System (Infections and infestations) | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Dengue Fever (Infections and infestations) | 1 | 0 | 0
Pericarditis Tuberculous (Infections and infestations) | 1 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Posterior Reversible Encephalitis Syndrome (Nervous system disorders) | 2 | 2 | 0
Intracranial Pressure Increased (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Cerebral Hemorrhage (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1
Congestive Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 0
Renal Failure Acute (Renal and urinary disorders) | 4 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Strangury (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Endocrine disorders) | 0 | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voclosporin Low Dose (N=89) | Voclosporin High Dose (N=88) | Placebo (N=88)
Glomerular Filtration Rate Decreased (Investigations) | 27 | 27 | 12
Diarrhoea (Gastrointestinal disorders) | 16 | 14 | 14
Nausea (Gastrointestinal disorders) | 16 | 11 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 5 | 3
Hypertension (Vascular disorders) | 15 | 14 | 8
Vomiting (Gastrointestinal disorders) | 15 | 9 | 10
Anaemia (Blood and lymphatic system disorders) | 13 | 14 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 18 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 12 | 9
Headache (Nervous system disorders) | 10 | 15 | 11
Oedema Peripheral (General disorders) | 9 | 7 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 5 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 4 | 2
Pyrexia (General disorders) | 6 | 9 | 1
Dyslipidamia (Metabolism and nutrition disorders) | 6 | 7 | 6
Urinary Tract Infection (Infections and infestations) | 6 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 6 | 6 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 7 | 5
Herpes Zoster (Infections and infestations) | 5 | 6 | 5
Nasopharyngitis (Infections and infestations) | 5 | 4 | 3
Gastroenteritis (Infections and infestations) | 5 | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3
Dizziness (Nervous system disorders) | 5 | 2 | 1
Insomnia (Psychiatric disorders) | 4 | 5 | 4
Gastroenteritis (Immune system disorders) | 5 | 3 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 3 | 7 | 0
Gingival Hypertrophy (Gastrointestinal disorders) | 3 | 6 | 0
Blood Pressure Increased (Investigations) | 3 | 5 | 1
Bronchitis (Infections and infestations) | 2 | 5 | 3
Oedema (General disorders) | 2 | 5 | 1
Tachycardia (Cardiac disorders) | 2 | 5 | 1
Oral Candidiasis (Infections and infestations) | 2 | 5 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 7 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No